CLINICAL TRIAL: NCT03702296
Title: Can the Use of Ear Plugs and Eye Masks Help to Improve Sleep Quality After Major Abdominal Surgery?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2018/2288
Record Dates: First submitted 2018-08-06; First posted 2018-10-11 (Actual); Last update posted 2019-10-14 (Actual); Status verified 2019-10

CONDITIONS: Sleep; Major Abdominal Surgery; Critical Care
MeSH Terms: interventions — Ear Protective Devices

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Blinded assessors will review the patients for 3 days post-operatively and assess sleep quality using the Richard-Campbell sleep questionnaire.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Other): Patients will be provided with ear plugs and eye masks, to be used from 10pm to 6am, for 3 days post-operatively.
  Interventions: Other: Ear plugs and eye masks
- Control (No Intervention): No ear plugs or eye masks provided.

INTERVENTIONS:
Other: Ear plugs and eye masks — Patients in the intervention arm will be provided with ear plugs and eye masks and instructed on the use of these during sleep
  Arms: Intervention

SUMMARY:
The importance of good sleep has been gaining interest in critically ill patients as poor sleep is associated with increased rates of delirium, non-invasive ventilation failure and stress to the patient.

The use of earplugs and eye masks has been shown to result in longer sleep time and better sleep quality. The primary outcome of this randomized control trial is to evaluate if the use of eye masks and earplugs in patients undergoing major abdominal surgery will lead to improved sleep quality. Secondary outcomes include the level of noise intensity in the various monitored units, incidence of delirium, nursing demand, length of hospitalization and anaesthetic techniques. With these findings, we hope to be able to improve patients' overall satisfaction with the healthcare received.

DETAILED DESCRIPTION:
The importance of good sleep has been gaining interest in critically ill patients as poor sleep has been found to be associated with increased rates of delirium, non-invasive ventilation failure, and may serve as a stressor to patients. The use of earplugs and eye masks to improve sleep quality has been described in the critically ill patient population and outcomes have suggested that such interventions have resulted in longer sleep time and Rapid Eye Movement sleep, shorter sleep onset latency and less awakenings, with an enhanced perceived sleep quality. In the post-anaesthesia care unit, these interventions have also led to significantly preserved sleep quality in patients. The primary outcome of this randomized control trial is to evaluate if the use of eye masks and earplugs in patients undergoing major abdominal surgery, and who will be admitted to a monitored unit postoperatively, will lead to improved sleep quality. Secondary outcomes evaluated include the level of noise intensity in the various monitored units (Intensive Care Unit/Intermediate Care Area/High Dependency Ward), incidence of delirium, nursing demand, length of hospitalization and anaesthetic techniques. With these findings, we hope to be able to improve patients' overall satisfaction with the healthcare received.

ELIGIBILITY:
Inclusion Criteria:

* All patients who are 21 years old and above, undergoing elective major abdominal surgery in Singapore General Hospital, and who are anticipated to require a monitored bed postoperatively will be identified via Operating Theatre Management system the day before surgery. Postoperatively, these patients must have a Glasgow Coma Scale of at least 10, able to obey verbal commands and stay in a monitored unit postoperatively (Intensive Care Unit/Intermediate Care Area/High Dependency).

Exclusion Criteria:

* Patients who have known hearing impairment, dementia, confusion, delirium or with a tracheostomy will be excluded.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-08-29 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-03-30 (Actual)

PRIMARY OUTCOMES:
Comparison of sleep quality between the 2 arms based on Richard Campbell sleep questionnaire | 3 days

SECONDARY OUTCOMES:
Comparison of overall patient satisfaction between the 2 arms based on Richard Campbell sleep questionnaire | 3 days
Frequency of nursing interventions required during the night | 3 days
  Subjective assessment by nurses
Incidence of delirium, based on twice daily scoring on the Neecham Confusion Tool | 3 days
  Neecham Confusion Tool consists of 9 scoring components: Attention (score of 0-4), Command (score of 0-5), Orientation (0-5), Appearance (0-2), Motor Behaviour (0-4), Verbal Behaviour (0-4), Vital Function Stability (0-2), Oxygen Saturation Stability (0-2) and Urinary Continence Control (0-2). The sum of the scores from each component is combined into a Total Neecham Score, with higher scores indicating that the patient is less likely at risk of delirium.
Duration of hospitalisation | through study completion, an average of 1 year
Noise intensity in the various monitored care units | 3 days
  Measured using a sound detector, in decibels

CONTACTS AND LOCATIONS:
Locations (1):
- Singapore General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Leong RW, Davies LJ, Fook-Chong S, Ng SY, Lee YL. Effect of the use of earplugs and eye masks on the quality of sleep after major abdominal surgery: a randomised controlled trial. Anaesthesia. 2021 Nov;76(11):1482-1491. doi: 10.1111/anae.15468. Epub 2021 Apr 21. PMID 33881774